CLINICAL TRIAL: NCT07304024
Title: A Double-Blinded, Placebo-Controlled, Randomized, Phase 1/2a Clinical Study to Test the Safety and Efficacy of a Treatment for a Form of Age-Related Central Auditory Processing Disorder Consisting of Clemastine Fumarate Plus Engineered Sound
Brief Title: A Treatment for a Form of Age-Related Central Auditory Processing Disorder Consisting of Clemastine Fumarate Plus Engineered Sound
Acronym: CAPD-LOOT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25-1184
Record Dates: First submitted 2025-12-19; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Central Auditory Processing Disorder; Hearing Impaired (Partially); Hearing; Hearing Abnormality; Hearing Disability; Hearing Disorder; Hearing Disorders; Hearing Impairment, Sensorineural; Hearing Handicap; Hearing Impaired; Hearing Impairment; Hearing Loss; Central Auditory Disease; Noise Exposure; Noise Induced Hearing Loss; Noise-Induced Hearing Loss; Sound Perception; Myelin Degeneration; Myelinopathy; Myelin Integrity; Remyelination; Hidden Hearing Loss; Cocktail Party Skill; Cocktail Party Syndrome; CAPD; Age Problem
Keywords: clemastine fumarate; Hidden Hearing Loss; Cocktail Party; Engineered Sound; Sound Therapy; central auditory processing disorder; Hearing in noise; oligodendrocyte; Localized Oligodendrocyte Optimization Therapy; LOOT; CAPD; Age-Related Hearing Loss
MeSH Terms: conditions — Language Development Disorders; Hearing Loss; Hearing Disorders; Hearing Loss, Sensorineural; Auditory Diseases, Central; Hearing Loss, Noise-Induced; Hearing Loss, Hidden; Presbycusis | interventions — Clemastine; Placebo Effect

STUDY DESIGN:
Intervention Model Description: Trial participants will be tested for hearing thresholds and ability to isolate a sound signal from background noise. If appropriate, they will then be enrolled into one of the four arms of the study and undergo the proposed one-month treatment. After the treatment period, participants will be tested again for hearing thresholds and their ability to isolate s sound source of interest from background noise.
  Adaptive parallel design with 4 initial arms. Interim analysis planned to assess whether the three control arms (placebo+sound, drug+white noise, placebo+white noise) show equivalent results as predicted by preclinical data. If confirmed, two control arms may be dropped to optimize study efficiency while maintaining scientific rigor.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study coordinators and all study personnel interacting with participants will be masked. The study statistician performing the interim analysis for the adaptive design will remain blinded to treatment allocation, using coded group assignments. A secondary statistician will evaluate study data as it is generated but will not have any contact with assigned participants or influence on study coordinators, care providers, or outcome assessors. Pharmacy staff preparing study medications will not be blinded but will have no participant contact.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Group (Experimental): Active clemastine fumarate + engineered sound stimulation
  Interventions: Combination Product: Clemastine Fumarate Combined With Engineered Sound
- Placebo Sound (Active Comparator): Active clemastine fumarate + placebo sound (white/pink noise)
  Interventions: Drug: Clemastine Fumarate Combined With Pink Noise
- Placebo Drug (Placebo Comparator): Placebo drug + engineered sound stimulation
  Interventions: Combination Product: Placebo Drug With Engineered Sound
- Control Group - Double Placebo (Placebo Comparator): Placebo drug + placebo sound (white/pink noise)
  Interventions: Combination Product: Placebo - Placebo

INTERVENTIONS:
Combination Product: Clemastine Fumarate Combined With Engineered Sound — Treatment Group:
  Drug: 16.08 mg clemastine fumarate (8.04 mg in the morning and 8.04 mg in the evening) during the first week of the 30 day treatment period, followed by 10.72 mg clemastine fumarate once daily in the evening for the remainder of the 30 day period. Tablets taken with water in morning and evening with or without food. This dosage corresponds to 12 mg clemastine base daily during the first week followed by 8 mg clemastine base daily for the remainder of the 30 day period. This matches dosing proven safe in previous Phase II multiple sclerosis trials.
  Sound: This medication will be combined with a proprietary engineered acoustic stimulus designed to activate central auditory processing pathways, delivered via provided headphones for 60 minutes daily during the 30-day treatment period. Sound consists of spatially modulated frequency sweeps targeting neural circuits involved in speech-in-noise processing. Participants instructed to listen during quiet, awake periods.
  Other Names: Localized Oligodendrocyte Optimization Therapy; LOOT
  Arms: Treatment Group
Drug: Clemastine Fumarate Combined With Pink Noise — Drug and Placebo Sound Group:
  Drug: 16.08 mg clemastine fumarate (8.04 mg in the morning and 8.04 mg in the evening) during the first week of the 30 day treatment period, followed by 10.72 mg clemastine fumarate once daily in the evening for the remainder of the 30 day period. Tablets taken with water in morning and evening with or without food. This dosage corresponds to 12 mg clemastine base daily during the first week followed by 8 mg clemastine base daily for the remainder of the 30 day period. This matches dosing proven safe in previous Phase II multiple sclerosis trials.
  Sound: Broadband white noise matched for average intensity to engineered sound. Delivered via provided headphones for 60 minutes daily during the 30-day treatment period. Serves as acoustic control to maintain participant and investigator blinding. Participants instructed to listen during quiet, awake periods.
  Other Names: Dayhist; Tavist
  Arms: Placebo Sound
Combination Product: Placebo Drug With Engineered Sound — Placebo Drug and Engineered Sound Group:
  Drug: Matching placebo tablets administered orally twice daily during the first week and once daily for the remainder of the 30 consecutive days. Tablets identical in appearance, taste, and smell to active drug. Taken with water in morning and evening with or without food.
  Sound: This placebo will be combined with a proprietary engineered acoustic stimulus designed to activate central auditory processing pathways, delivered via provided headphones for 60 minutes daily during the 30-day treatment period. Sound consists of spatially modulated frequency sweeps targeting neural circuits involved in speech-in-noise processing. Participants instructed to listen during quiet, awake periods.
  Arms: Placebo Drug
Combination Product: Placebo - Placebo — Placebo Drug and Placebo Sound Group:
  Drug: Matching placebo tablets administered orally twice daily during the first week and once daily for the remainder of the 30 consecutive days. Tablets identical in appearance, taste, and smell to active drug. Taken with water in morning and evening with or without food.
  Sound: Broadband white noise matched for average intensity to engineered sound. Delivered via provided headphones for 60 minutes daily during the 30-day treatment period. Serves as acoustic control to maintain participant and investigator blinding. Participants instructed to listen during quiet, awake periods.
  Arms: Control Group - Double Placebo

SUMMARY:
The goal of this clinical trial is to determine the efficacy of Clemastine Fumarate in the presence of engineered sound to treat age-related central auditory processing disorder (CAPD). This disorder impacts 800M patients worldwide, including ~1/3 people over 40 years of age and ~1/2 people over 65, resulting in an inability to hear in noisy environments.

The primary hypothesis this study aims to test is: engineered sound, driving localized neural circuit activity, will enable Clemastine Fumarate to mature Oligodendrocyte cells and thus remyelinate these activated neural circuits. This Localized Oligodendrocyte Optimization Therapy (LOOT) was highly effective in preclinical animal studies so this clinical trial aims to answer if this therapy will translate to humans.

The study is an adaptive design intended to compare the efficacy of the drug in the presence or absence of the engineered sound for improving hearing in noise ability. Trial participants will be tested for hearing thresholds and ability to isolate a sound signal from background noise. If they meet the inclusion criteria, they will be enrolled into one of the four arms of the study and undergo the proposed one-month treatment (drug and sound or respective placebos). After the treatment period, trial participants will be tested again for hearing thresholds and their ability to isolate s sound source of interest from background noise. The hypothesis to be tested in this clinical trial is that the one-month treatment will significantly improve the participant's ability to isolate a sound source of interest from background noise.

The design has four arms, drug+sound, placebo+sound, drug+white noise, and placebo+white noise. Based on our preclinical data, control arms are all expected to show identical results, thus our adaptive design includes interim analyses to allow for dropping of two of the three placebo arms should the preclinical results be replicated as anticipated.

We will also monitor each participant's general health during the duration of the clinical trial, which will be done by performing a number of blood tests, an EKG and a general physical before and after the one-month treatment period. We expect no significant changes since participants will take the drug for the one-month period at dosages already demonstrated safe in several Phase II studies of multiple sclerosis. Similarly, the engineered sound will be listened to for one hour per day during this month at sound intensities well below threshold that might cause noise-induced hearing damage.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 45 and 65 years old (middle aged) at the screening/enrollment visit (Visit 1).
* Written informed consent obtained from the subject and ability for the subject to comply with the requirements of the study.
* Documentation of no more than a mild high-frequency hearing sensitivity loss and normal middle-ear function will be obtained using standard audiometric equipment with measurements done by an audiologist; Specifically, testing will show:

  * bilateral hearing thresholds < 20 dB HL at audiometric frequencies from 250 Hz to 4000 Hz inclusively, with no air-bone gaps > 10 dB.
  * symmetrical hearing thresholds between the ears through 8000 Hz, defined as <20 dB difference at any single audiometric frequency or < 15 dB difference at 2 or more contiguous frequencies.
  * normal (Type A) tympanograms bilaterally.
* No cognitive deficit shown upon screening with the Montreal Cognitive Assessment (MOCA) test (Nasreddine et al. 2005).
* Distortion product otoacoustic emission (DPOAE) showing no more than 20 dB hearing loss at audiometric frequencies from 250 Hz to 4000 Hz.
* Subjects failing the hearing in noise test at 15 degrees. Failing is defined as SNR being 12 dB below from what is found in normal hearing subjects without central hearing loss.

Exclusion Criteria:

* Any subjects who do not fall under the criteria defined above.
* Any of the following conditions which are listed as contraindications or warnings for use of the clinical trial drug (from labeling):

  * Known sensitivity to clemastine fumarate or other antihistamines of similar composition
  * Pregnancy or nursing mother as determined objectively with a urine pregnancy test
  * Lower respiratory tract disease including asthma, or breathing difficulties such as emphysema or chronic bronchitis
  * Glaucoma or increased intraocular pressure
  * Stenosing peptic ulcers or pyloroduodenal obstruction
  * Trouble urinating due to an enlarged prostate gland. Mild urinary issues (Stage 1 Benign Prostatic Hyperplasia) will not be considered an automatic exclusion but it must be emphasized to patients with this diagnosis that difficulty urinating is a possible side effect that may compound their BPH symptoms.
  * Significant cardiovascular disease, chronic hypertension or hypotension
  * Hyperthyroidism
  * Alcoholism- as defined by consuming on average 3+ drinks per day for women or 4+ drinks per day for men or previous diagnosis of alcohol use disorder by a clinician as defined by DSM V criteria.
  * Patients with a history of seizures will be excluded.
  * Patients with evidence of suicidal ideation/behavior as assessed by the Columbia Suicide Severity Rating Scale (C-SSRS).
* We will generally exclude subjects with significant or uncontrolled medical disorders (e.g., hepatic, hematologic, renal, gastrointestinal, neurological, psychiatric disorders). We will define these patients as those who fall outside of normal ranges for a physical examination of vital signs, a 12-lead EKG, and a safety clinical laboratory assessment including complete blood count (CBC) and comprehensive metabolic panel (CMP). Exclusion with these tests will specifically focus on identifying the following disorders based on the listed criteria:
* Leukopenia as defined as a CBC white blood cell count < 4000/ul
* Anemia as defined by a CBC Hemoglobin <9.0 g/dL or <10.0 g/dL (Grade 2+ CTCAE)
* Lymphopenia as defined by CBC Absolute lymphocyte count <1000/µL.
* Neutropenia as defined by CBC ANC <1500/µL (solid tumors), ANC <1000/µL (hematologic malignancies). In the case of participants with African, Middle Eastern or West Indian descent a clinician's judgement will be considered to assess the possibility of benign ethnic neutropenia which is not an exclusion criteria.
* Thrombocytopenia as defined by CBC Platelet count <75000/µL
* Hepatic Impairment based on CMP: Total bilirubin >1.5× ULN, AST/ALT >3× ULN (or >5× ULN if liver metastases), Alkaline phosphatase >3× ULN.
* Hepatic Impairment based on CMP: Serum creatinine >2.0 mg/dL (alternative threshold).
* Metabolic abnormalities based on CMP: Albumin <3.0 g/dL
* Taking medications that would contraindicate taking the clinical trial drug; Specifically, (from labeling):

  * Monoamine oxidase inhibitor therapy
  * CNS depressants (sedatives, tranquilizers, hypnotics)
* A history of significant otologic disorder such as repetitive ear infections or Meniere's disease
* A history of significant neurologic disorder, or current neurodegenerative diseases such as multiple sclerosis, which could present a confound and impact the electrophysiological outcome measures.
* A history of traumatic brain or closed head injury because this can cause symptoms of central auditory processing problems unrelated to aging and demyelination.
* English as a second language (non-native English speakers), which is known to negatively impact scores on speech recognition testing.
* Presence of any other condition or abnormality that in the opinion of the Investigator or his co-PIs would compromise the safety of the patient or the quality of the data.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Improvement in hearing-in-noise at 15 degree separation | At enrollment and again after intervention (Week 5 or 6)
  Measures ability to understand speech in background noise, tested in a sound chamber with speakers arranged in a circle. Participants listen to sentences spoken by a female speaker while 6-person babble noise plays from a speaker 15 degrees away. Test uses Harvard IEEE sentences (5 keywords each) at 60 dB with varying signal-to-noise ratios (SNR). Participants repeat words they hear. An adaptive procedure determines the SNR needed for 40% accuracy (>2/5 words correct) and 80% accuracy (>4/5 words correct). Lower SNR values indicate better performance. Primary outcome is change in SNR from baseline to post-treatment (Day 30). This tests central auditory processing, not peripheral hearing, as it requires the brain to separate speech from noise when sounds come from different directions. Analysis uses linear regression comparing treatment groups to placebo for change in SNR, with p<0.017 considered significant due to multiple endpoints. Success is group-wise improvement of >3dB.
Improvement in hearing-in-noise at 30 degree separation | At enrollment and again after intervention (Week 5 or 6)
  Measures ability to understand speech in background noise, tested in a sound chamber with speakers arranged in a circle. Participants listen to sentences spoken by a female speaker while 6-person babble noise plays from a speaker 30 degrees away. Test uses Harvard IEEE sentences (5 keywords each) at 60 dB with varying signal-to-noise ratios (SNR). Participants repeat words they hear. An adaptive procedure determines the SNR needed for 40% accuracy (>2/5 words correct) and 80% accuracy (>4/5 words correct). Lower SNR values indicate better performance. Primary outcome is change in SNR from baseline to post-treatment (Day 30). This tests central auditory processing, not peripheral hearing, as it requires the brain to separate speech from noise when sounds come from different directions. Analysis uses linear regression comparing treatment groups to placebo for change in SNR, with p<0.017 considered significant due to multiple endpoints. Success is group-wise improvement of >3dB.

SECONDARY OUTCOMES:
Speech, Spatial, and Qualities questionnaire (SSQ) | At enrollment and again after intervention (Week 5 or 6)
  Speech, Spatial, and Qualities questionnaire (SSQ) by Gatehouse & Noble, 2004. Self-report questionnaire assessing speech understanding, spatial hearing, and sound quality in daily life. The evaluation ranges from 0-10 for each item. With higher scores indicating better function.
Tinnitus Handicap Inventory [THI] | At enrollment and again after intervention (Week 5 or 6)
  Newman et al., 1996. 25-item questionnaire measuring tinnitus severity and impact on daily life. Scores range from 0-100 with higher scores indicating greater handicap.
Wave III amplitude of the ABR | At enrollment and again after intervention (Week 5 or 6)
  This physiological measurement is not relevant in the participant's daily life, however, changes in ABR waves will give us valuable insights into the mechanisms of the treatment. ABR will be measured via existing predicate devices and/or with FDA cleared EEG devices and standard auditory stimuli appropriate for measuring auditory brainstem response (ABR) waves. This assessment is non-invasive and involves an electrode placed on appropriate locations of a participants head to record electrophysiologic activity while the patient listens to auditory stimuli such as clicking that stimulates the relevant neural circuits.

OTHER OUTCOMES:
Audiological Safety & Eligibility | At enrollment and again after intervention (Week 5 or 6)
  Auditory function assessments will include: Audiogram, and Distortion product otoacoustic emission (DPOAE) tests. For the audiogram and DPOAE, right, left, and bilateral thresholds will be recorded in the range of 250-8000 Hz. To include subjects or determine if an adverse event (AE) has occured, these measures will verify normal thresholds and symmetrical hearing between the ears. On the bilateral audiogram the normal threshold is < 21 dB hearing loss in the range of (250-4000 Hz) and no air-bone gaps >10 dB. Symmetrical hearing will be defined by <21 dB differences OR any single frequency and <16 dB difference at 2+ contiguous frequencies. For the DPOAE <20 dB hearing loss will be defined as normal. Clinician judgement will be used to over-rule exclusion or determination of AE.
Participant Journal | Journal entries will be recorded daily during intervention and returned upon final evaluation (Week 5 or 6)
  A participant journal will be completed during the trial to assess deviations from compliance or other self-reported observations.

CONTACTS AND LOCATIONS:
Overall Officials: Achim Klug, PhD, Principal Investigator — Colorado University Anschutz Medical Center; Samuel A Budoff, PhD, MS, Study Director — Colorado University Anschutz Medical Center
Locations (1):
- University of Colorado Anschutz Medical Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to: (1) proprietary nature of the engineered acoustic intervention which is core intellectual property, (2) potentially small sample size due to potential early stopping creates re-identification risks despite de-identification efforts, and (3) lack of dedicated data sharing infrastructure as an academic investigator led trial. Aggregate results will be published in peer-reviewed journals.

REFERENCES:
- [Background] Green AJ, Gelfand JM, Cree BA, Bevan C, Boscardin WJ, Mei F, Inman J, Arnow S, Devereux M, Abounasr A, Nobuta H, Zhu A, Friessen M, Gerona R, von Budingen HC, Henry RG, Hauser SL, Chan JR. Clemastine fumarate as a remyelinating therapy for multiple sclerosis (ReBUILD): a randomised, controlled, double-blind, crossover trial. Lancet. 2017 Dec 2;390(10111):2481-2489. doi: 10.1016/S0140-6736(17)32346-2. Epub 2017 Oct 10. PMID 29029896
- [Background] Mei F, Fancy SPJ, Shen YA, Niu J, Zhao C, Presley B, Miao E, Lee S, Mayoral SR, Redmond SA, Etxeberria A, Xiao L, Franklin RJM, Green A, Hauser SL, Chan JR. Micropillar arrays as a high-throughput screening platform for therapeutics in multiple sclerosis. Nat Med. 2014 Aug;20(8):954-960. doi: 10.1038/nm.3618. Epub 2014 Jul 6. PMID 24997607
- [Background] Manousi A, Kury P. Small molecule screening as an approach to encounter inefficient myelin repair. Curr Opin Pharmacol. 2021 Dec;61:127-135. doi: 10.1016/j.coph.2021.09.008. Epub 2021 Nov 6. PMID 34753035
- [Background] Schran HF, Petryk L, Chang CT, O'Connor R, Gelbert MB. The pharmacokinetics and bioavailability of clemastine and phenylpropanolamine in single-component and combination formulations. J Clin Pharmacol. 1996 Oct;36(10):911-22. doi: 10.1002/j.1552-4604.1996.tb04758.x. PMID 8930778
- [Background] Cox RM, Alexander GC, Gilmore C. Development of the Connected Speech Test (CST). Ear Hear. 1987 Oct;8(5 Suppl):119S-126S. doi: 10.1097/00003446-198710001-00010. PMID 3678650
- [Background] Gatehouse S, Noble W. The Speech, Spatial and Qualities of Hearing Scale (SSQ). Int J Audiol. 2004 Feb;43(2):85-99. doi: 10.1080/14992020400050014. PMID 15035561
- [Background] Killion MC, Niquette PA, Gudmundsen GI, Revit LJ, Banerjee S. Development of a quick speech-in-noise test for measuring signal-to-noise ratio loss in normal-hearing and hearing-impaired listeners. J Acoust Soc Am. 2004 Oct;116(4 Pt 1):2395-405. doi: 10.1121/1.1784440. PMID 15532670
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Newman CW, Jacobson GP, Spitzer JB. Development of the Tinnitus Handicap Inventory. Arch Otolaryngol Head Neck Surg. 1996 Feb;122(2):143-8. doi: 10.1001/archotol.1996.01890140029007. PMID 8630207